CLINICAL TRIAL: NCT05466786
Title: Landscape Ofhomologous Recombination-related (HRR) Genes Mutations and HRD, and Correlation With Survival in HER2-lowbreast Cance
Brief Title: Distribution of the Homologous Recombination-related (HRR) Genesmutationsand HRD in Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chang Gong, Chief physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2022-030-01
Record Dates: First submitted 2022-07-10; First posted 2022-07-20 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; HER2-low Breast Cancer
Keywords: Homologous recombination-related; Homologous recombination deficiency
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Sample Name：blood Note：Return any surplus after use
  2. Sample Name：Tumor tissue Note：Return any surplus after use
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental ARM: All patients received standard care for postoperative management.
  Interventions: Other: Standard Management

INTERVENTIONS:
Other: Standard Management — Standard Management

SUMMARY:
This is a cross-sectional and an observational study, investigator-initiated study in HER2-low breast cancer patients. Approximately 255 subjects with HRD (homologous recombination deficiency) assessment will be enrolled in this study to examine the distribution and features of HRD/HRR (homologous recombination repair).

In this study, investigators plan to clarify the frequency of HRR/HRD in Chinese patients with HER2-low breast cancer.

In addition, it is planned to investigate any association between invasive disease-free survival (iDFS)/overall survival (OS) and HRD/HRR in HER2-low breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-70 years with pathologically confirmed HER2-low breast cancer (defined as IHC 2+/ISH- or IHC 1+ per ASCO/CAP guidelines);
2. ECOG performance status of 0 or 1;
3. Treatment-naïve operable primary breast cancer with completed homologous recombination deficiency (HRD) assessment;

5）Absence of distant metastasis; 6）Availability of adequate tumor tissue and blood samples for biomarker analysis.

Exclusion Criteria:

1. Recurrent or inoperable locally advanced breast cancer;
2. Bilateral breast cancer;
3. History of other malignant tumors within the past 5 years;
4. Incomplete clinical or pathological data.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients aged 18-70 years with pathologically confirmed HER2-low breast cancer (defined as IHC 2+/ISH- or IHC 1+ per ASCO/CAP guidelines)
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2022-08-07 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
1.To assess the distribution characteristics of mHRR/HRD in breast cancer with low HRE2 expression in Chinese population | At the time of 4 weeks after surgery
  the distribution and features of HRD /HRR is evaluated.

SECONDARY OUTCOMES:
To assess the clinical characteristics between patients with mutations and non-mutation | At the time of 4 weeks after surgery
  Association between mutations and non-mutations group in HRD/HRR is assessed.
To compare the correlation between iDFS/OS and different adjuvant treatment regimens for breast cancer with low HER2 expression | At the time of 36 months after surgery
  IDFS, was a composite endpoint defined as the time from enrollment until the date of the first occurrence of one of the following events: Ipsilateral invasive breast cancer recurrence (same breast); Ipsilateral (same side of body) local regional invasive breast cancer recurrence (axilla, regional lymph nodes, chest wall, and/or skin); Distant recurrence (evidence of breast cancer in any anatomic site); Death attributable to any cause; Contralateral (opposite side of the body) invasive breast cancer.
  3-year Overall survival (OS) was defined as time from date of randomization to death from any cause, otherwise cases were censored at date last known to be alive.
  Association between IDFS/OS and HRD/HRR information is evaluated.
To investigate the HRR/HRD characteristics and clinical characteristics (family history, age pathological feature es, etc.) of breast cancer patients with low HER2 expression | At the time of 4 weeks after surgery
  Association between multivariate prognostic factors and survival is evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Gong Chang, doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No